CLINICAL TRIAL: NCT04691271
Title: Effect of Early Stellate Ganglion Block for Cerebral Vasospasm After Aneurysmal Subarachnoid Hemorrhage: a Randomized Controlled Trial (BLOCK-CVS)
Brief Title: Stellate Ganglion Block and Cerebral Vasospasm
Acronym: BLOCK-CVS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Z191100006619068
Record Dates: First submitted 2020-12-13; First posted 2020-12-31 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-01

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Stellate Ganglion Block; Cerebral Vasospasm
Keywords: Cerebral vasospasm; Stellate ganglion block
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In addition to routine anesthesia management and surgical operations, a stellate ganglion block was performed before induction of anesthesia, and then receive standard care after operation. Related statistical indicators were collected prospectively.
  Interventions: Procedure: Stellate ganglion block
- Blank control group (No Intervention): In this study, a blank control was used. Routine anesthesia management and surgical operation were used without any special interventions(only an camouflaging action), and then receive standard care after operation. Only relevant statistical indicators were collected prospectively.

INTERVENTIONS:
Procedure: Stellate ganglion block — After the patient entered the operating room, early SGB will be performed by a designated experienced anesthesiologist using the B-ultrasound visualization technique. The intervention site is the ipsilateral side of the planned craniotomy site. After routine disinfection, 0.5% ropivacaine 8-10 mL will be injected into the surface of the longus colli muscle on the medial side of the prevertebral fascia at the level of the C6 anterior tubercle, and then the puncture point will be covered with sterile dressings. The success criteria of e-SGB are Horner's syndrome, which is characterized by a miosis, ptosis, enophthalmos, conjunctival hyperemia and facial reddishness without sweating. For the "camouflaging" arm, the anesthesiologist only covered the corresponding part of the patient with sterile dressings to confuse the follow-up, without any puncture. All patients will be admitted to the ICU after the operation and then receive the standard of care.
  Arms: Intervention group

SUMMARY:
At present, cerebral vasospasm (cVS) is the main cause of delayed cerebral infarction (DCI), which leads to high disability and mortality rate after aneurysmal subarachnoid hemorrhage. As a consequence, the key of reducing DCI is to prevent cVS. But unfortunately, despite years of efforts, the prevention and treatment of cVS is still a major clinical dilemma and various ways of treatment are still being explored. Recent studies have shown that stellate ganglion block (SGB) can dilate cerebral vessels and alleviate the impact of existing cVS. However, there is no study to evaluate the effect of early application of SGB on the improvement and prevention of cVS after aSAH.

DETAILED DESCRIPTION:
Cerebral vasospasm refers to the extensive segmental or diffuse contraction of cerebral vasculature after aSAH, and cerebral blood flow is significantly reduced, which can lead to delayed cerebral ischemia (DCI) or delayed ischemic neurological dysfunction (DIND). Past studies have shown that if cerebral vasospasm occurs in patients with aSAH, the proportion of ischemic brain injury can be as high as 20%-30%.Obviously, prevention and treatment of CVS are the key to reducing the disability and mortality of aSAH.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-65 years old;
* Within 48 hours after onset of aSAH,and planning surgical treatment(aneurysm clipping);
* Preoperative Hunt-Hess grade 2-3
* Sign informed consent.

Exclusion Criteria:

* ASA > grade III;
* Patients with posterior circulation aneurysm, ophthalmic aneurysms or internal carotid aneurysms;
* patients with multiple aneurysms;
* Patients with severe coagulation dysfunction;
* Patients with trauma and local infection in the nerve block area;
* Local anatomic structure changes (neck structure changes caused by radiotherapy, chemotherapy and surgery);
* MCA stenosis or infarction was found by preoperative imaging;
* Patients with poor temporal window signal revealed by preoperative TCD (clear waveform image could not be obtained);
* Allergy to known local anesthetics;
* Pregnant and lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of symptomatic vasospasm during hospitalization | an average of 2 weeks
  Symptomatic vasospasm is defined as new focal or global neurological dysfunction or a decrease in the Glasgow coma score by more than 2 points, and with angiographic vasospasm on TCD or CTA.

SECONDARY OUTCOMES:
The incidence of TCD vasospasm during hospitalization | on the days 3-5 after operation
  The mean blood flow velocity (MFV) of the middle cerebral artery ≥ 120 cm/s or Lindegaard index (ratio of MFV of the middle cerebral artery to the internal carotid artery) ≥ 3.
The incidence of CTA vasospasm on the days 3-5 after operation | on the days 3-5 after operation
  Compared with the preoperative baseline, the corresponding vessel diameter narrowed by more than 30% or new segmental stenosis occurred, not related to atherosclerosis or mechanical artery stenosis caused by arterial clamps or coils.
The incidence of hypoperfusion in CTP diagnosis on the days 3-5 after operation | on the days 3-5 after operation
  The incidence of hypoperfusion in CTP diagnosis
The incidence of new cerebral infarction observed on the days 90 after operation and discharge . | on the days 90 after operation and discharge
  New cerebral infarction is defined only as the appearance of new low-density infarct shadow on CT image compared with preoperation.
The changes of he mean blood flow velocity (mBFV) after operation | on the days 3-5 after operation
  the changes in the mean blood flow velocity (mBFV) of all large intracranial anterior circulation vessels
Total length of stay in the intensive care unit and hospital. | on the 90 days
  Days
The modified Rankin scale at discharge, 30days, and 90 days | on the 30 and 90 days
  The modified Rankin scale ≤2 is defined as good prognosis
All-cause mortality rate up to 90 days. | on the 90 days
  The rate
Postoperative delirium incidence during hospitalization | on the days 1-3 after operation
  The rate
Postoperative cognitive dysfunction | At discharge，an average of 2 weeks
  The rate
The proportion of remedial treatment after CVS | At discharge，an average of 2 weeks
  The rate
Adverse events during hospitalization | At discharge，an average of 2 weeks
  Myocardial infarction, cardiac arrest, pulmonary embolism, infection, SGB related complications, etc

CONTACTS AND LOCATIONS:
Overall Officials: Ruquan Han, M.D., Ph.D, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wu Y, Lin F, Bai Y, Liang F, Wang X, Wang B, Jian M, Wang Y, Liu H, Wang A, Chen X, Han R. Early stellate ganglion block for improvement of postoperative cerebral blood flow velocity after aneurysmal subarachnoid hemorrhage: results of a pilot randomized controlled trial. J Neurosurg. 2023 Apr 28;139(5):1339-1347. doi: 10.3171/2023.3.JNS222567. Print 2023 Nov 1. PMID 37119094
- [Derived] Jing L, Wu Y, Liang F, Jian M, Bai Y, Wang Y, Liu H, Wang A, Chen X, Han R. Effect of early stellate ganglion block in cerebral vasospasm after aneurysmal subarachnoid hemorrhage (BLOCK-CVS): study protocol for a randomized controlled trial. Trials. 2022 Nov 4;23(1):922. doi: 10.1186/s13063-022-06867-9. PMID 36333751